CLINICAL TRIAL: NCT04730180
Title: Evaluating the Effectiveness of Different Targeting Approaches for Transcranial Magnetic Stimulation Treatment of Depression
Brief Title: Comparison of Targeting Methods for Transcranial Magnetic Stimulation Treatment of Depression
Acronym: XRnav
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer McNab, Associate Professor of Radiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60006
Record Dates: First submitted 2021-01-21; First posted 2021-01-29 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- No neuronavigation (Active Comparator): For this group, the stimulation location for repetitive transcranial stimulation treatment is estimated by the clinician via scalp measurements.
  Interventions: Device: Transcranial Magnetic Simulation
- Mixed reality neuronavigation (Active Comparator): For this group, the stimulation location for repetitive transcranial stimulation treatment is estimated by the clinician via a mixed reality neuronavigation device.
  Interventions: Device: Transcranial Magnetic Simulation; Device: Mixed reality neuronavigation

INTERVENTIONS:
Device: Transcranial Magnetic Simulation — Brain stimulation treatment will be performed using FDA-cleared TMS coils according to their intended use of treatment of medication resistant depression by targeting the dorsolateral prefrontal cortex.
Device: Mixed reality neuronavigation — Targeting of the dorsolateral prefrontal cortex will be performed with the help of a mixed reality neuronavigation system.
  Arms: Mixed reality neuronavigation

SUMMARY:
We aim to learn whether use of a mixed reality device for transcranial magnetic stimulation (TMS) targeting can improve treatment outcomes compared to targeting through scalp measurements or a commercial neuronavigation system. Prior studies indicate that neuronavigation can lead to improved treatment outcomes compared to scalp measurements, but neuronavigation adaption has been lacking due to the increased burden of the neuronavigation setup on the TMS operator. We will assess whether use of a mixed reality device can decrease that burden and speed up the neuronavigation process and is feasible to be used in a clinical setting.

DETAILED DESCRIPTION:
Prior studies suggest that treatment efficacy for TMS treatment of depression is affected by the targeting method used to guide TMS coil placement. We will compare the treatment outcome for three patient groups. TMS coil placement is guided for group 1) with simple scalp measurement targeting, for group 2) with a mixed reality neuronavigation system.

The treatment schedule for the medically prescribed TMS treatment for each patient are 30 daily weekday repetitive TMS treatments for 6 weeks with an additional 6 treatments tapered over 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ages 18-75.
2. MRI scanning eligibility, including no evidence of any form of metal embedded in the body (e.g., metal wires, nuts, bolts, screws, plates, sutures), as these produce artifacts when brain imaging. All potential subjects for the MRI component will need to successfully complete the screening forms at the Stanford Center for Cognitive and Neurobiological Imaging (CNI) or the Lucas Center. Those subjects who present no contraindications to being scanned will be allowed to participate.
3. Healthy subjects with no history of any Axis I psychiatric disorder, are taking psychotropic medication, or use illicit drugs.
4. Clinical subjects with a diagnosis of treatment resistant depression and prescribed a clinical course of treatment with rTMS.

Exclusion Criteria:

1. Any contraindication to being scanned in the 3.0T scanner at the Lucas Center or CNI such as having a pacemaker or implanted device that has not been cleared for scanning at 3.0 Tesla.
2. History of neurological disorders including but not limited to brain surgery, deep brain stimulation, radiation treatment, brain hemorrhage or tumor, stroke, seizures or epilepsy, head trauma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with response to TMS | 9 weeks
  We will count how many participants responded to TMS treatment in each arm. Response is measured as a more than 50% reduction in MADRS score per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A McNab, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No